CLINICAL TRIAL: NCT00286676
Title: The Use of Nutropin Depot in HIV-infected Adult Males
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-045
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Human Growth Hormone; Glucose Tolerance Test; Absorptiometry, Photon

INTERVENTIONS:
Drug: Nutropin
Procedure: Oral Glucose Tolerance Test
Procedure: Dual Energy X-ray Absorptiometry (DEXA)
Procedure: Computed Tomography (CT) Scan

SUMMARY:
This is a pilot study. We will treat 10 HIV-infected adults (1/2 with lipoatrophy) with GH depot for one year. Results will be compared to data from 10 HIV patients (1/2 with lipoatrophy), treated with Nutropin AQ subcutaneously. The primary endpoint of the study is to determine the effect of GH depot on body weight and lean tissue mass (LTM).

The secondary endpoints are to document changes in: 1) whole body protein turnover (WBPT), 2) gluconeogenesis, 3) bone mineral density and markers of bone turnover, 4) fat distribution (lipoatrophy), 5) thymus size, 6) T-cell subsets, and 7) TNF-µ levels. Adverse events, such as glucose intolerance and edema, will be monitored at every visit.

DETAILED DESCRIPTION:
Patients will be recruited from the HIV clinics at University of Texas Southwestern Medical School and the Veterans Administration Hospital by direct invitation from Dr. Margolis (adult HIV clinic director and University director for the NIH-ACTG). We will recruit 20 HIV-infected adult males who have been treated with stable protease inhibitor therapy regimen for the past 6 months. One half of the subjects will have evidence of lipoatrophy (as defined by the ACTG29). Each subject will have baseline (BL) measures made, and then will start on GH depot or subcutaneous AQ. Patients will be followed every two weeks for the first six weeks, then every three months for the remainder of the study. Study parameters to be measured include (also see flow chart in appendix):

* Baseline, 3, 6 and 12 months: OGTT, testosterone level, whole body protein turnover, hepatic glucose production and gluconeogenesis measures, DXA scan (for measuring lean tissue mass and bone density), bone mineral markers, resting energy expenditure, calorie count, T cell subsets, TNF µ levels.
* Every 3 months: IGF-1 (will obtain every 2 weeks for first 6 weeks), body weight, and post-prandial glucose level.
* Baseline, 6 and 12 months- CT scan for measurement of thymus size

ELIGIBILITY:
Inclusion Criteria:

* adult males ≥ 18 years of age
* mild to moderate lipoatrophy
* stable protease inhibitor therapy for at least six months.

Exclusion Criteria:

* Con-current supra-infection with acute illness defined by fever or bacterial culture
* malignancy
* females
* diabetes mellitus
* CNS tumors.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02-01 (Estimated); Primary Completion 2006-02-01 (Estimated); Study Completion 2006-02-01 (Estimated)

PRIMARY OUTCOMES:
1) body weight
2) lean tissue mass (LTM).
Testosterone levels

SECONDARY OUTCOMES:
1) whole body protein turnover (WBPT)
2) gluconeogenesis
3) bone mineral density and markers of bone turnover
4) fat distribution (lipoatrophy)
5) thymus size
6) T-cell subsets
7) TNF-µ level

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (3):
- United States (3):
  - Aston Ambulatory Care Center, Dallas, Texas
  - Parkland Health & Hospital System, Dallas, Texas
  - Veteran's Affairs Medical Center, Dallas, Texas